CLINICAL TRIAL: NCT03449693
Title: Efficacy of Oral Supplementation With Magnesium to Reduce Febrile Neutropenia in Pediatric Oncology Patients Treated With Cisplatin-Based Chemotherapy: Randomized Clinical Trial
Brief Title: Efficacy of Oral Supplementation With Magnesium to Reduce Febrile Neutropenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Collaborators: Hospital Infantil de Mexico Federico Gomez (Other); Centro de Investigación y Estudios Avanzados del Instituto Politécnico Nacional (Unknown)
Responsible Party: Principal Investigator, Osvaldo Daniel Castelan Martinez, Full Time Associate Professor C, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIM-2017-085
Record Dates: First submitted 2018-02-21; First posted 2018-02-28 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Febrile Neutropenia
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Intervention Model Description: Two groups: Intervention group and control group. The intervention group will receive institutional care protocol plus oral supplementation with magnesium. The control group will receive institutional care protocol only.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Magnesium Oxide Supplement (Experimental): Magnesium Oxide 250 mg tablet, daily for 30 days.
  Interventions: Dietary Supplement: Magnesium Oxide Supplement
- No Supplement (No Intervention): No Intervention

INTERVENTIONS:
Dietary Supplement: Magnesium Oxide Supplement — Magnesium Oxide tablet
  Other Names: M250
  Arms: Magnesium Oxide Supplement

SUMMARY:
Clinical Trial. Open label. Parallel Groups. The purpose of the study is to determine the efficacy of oral supplementation with magnesium oxide to reduce febrile neutropenia episodes in pediatric oncology patients treated with cisplatin-based chemotherapy.

DETAILED DESCRIPTION:
Febrile neutropenia (FN) is a worrying outcome in children receiving chemotherapy because it increments the risk of major complications, reduces quality of life and increments treatment costs. Moreover, it is the most common diagnosis in pediatric oncology patients that enter emergency rooms and the second most important cause of hospitalization, just behind hospitalization for administration of chemotherapy.

In Mexico, incidence of FN is of 62% of children with solid tumors treated with cisplatin-based chemotherapy (CBC). Cisplatin is one of the most nephrotoxic drugs being used in clinical settlements. The assessment of nephrotoxicity is made with the manifestation of tubular damage that causes electrolyte losses, specially of magnesium. Recently, our investigation group reported that there is an association of hypomagnesemia and the apparition of FN. This association has a biologic explanation in the fact that magnesium is a necessary cofactor for the neutrophil's diapedesis and the activation of complement cascade. To our knowledge, the role of magnesium supplementation has not been explored. With this evidence in mind, the investigators wondered if oral supplementation with magnesium will reduce FN episodes in pediatric oncology patients treated with CBC.

Objective: Determine the efficacy of oral supplementation with magnesium to reduce FN episodes in pediatric oncology patients treated with CBC.

Hypothesis: Previous clinical trials made in adult population have reported that supplementation with magnesium salts reduce episodes of hypomagnesemia in between 13 and 50%. Thus, oral supplementation with magnesium oxide will reduce 20% of FN episodes in pediatric oncology patients treated with CBC.

Materials and Methods: Randomized Clinical Trial, open-label, parallel groups of children over the age of nine with solid tumors treated with CBC at the Haemato-Oncology Department of the Hospital Infantil de México. To prove the hypothesis, it is required to randomize 107 CBC cycles to the intervention group and 107 CBC cycles to the control group. The sample size calculation was made by using the two proportions formula. Randomize of children will be made when they receive CBC indication. Patients assigned to the intervention group will receive institutional attention protocol plus a bottle of magnesium oxide, at the moment of hospitalization discharge. Patients assigned to the control group will receive only institutional attention protocol. The follow-up of patients will be made until an episode of FN appears or until the patient comes back for another CBC cycle. FN assessment will be measured with a unique temperature >38.3°C or a sustained temperature >38°C over the course of an hour plus a count of neutrophils under 1000 cells/mm3. The efficacy of oral supplementation with magnesium oxide will be determined by a Relative Risks calculation with confidence interval of 95% (CI95%). Moreover, Absolute Risk Reduction will be calculated, as well as Necessary Number to Treat. To adjust the principal variable a multivariate analysis will be made with a multiple logistic regression. The analysis will be made by protocol and by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients > 9 years old
* Pediatric patients with solid tumors treated with cisplatin-based chemotherapy
* Signing of Informed Consent from the parents
* Signing of Informed Assent from the children

Non-inclusion Criteria:

* Patients whose parents do not sign the Informed Consent
* Patients with magnesium losing tubulopathy
* Patients with hypomagnesemia previous to the cisplatin-based chemotherapy

Exclusion Criteria:

- Patients whose parents retire the Informed Consent

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 214 (Estimated)
Dates: Start 2017-10-19 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Febrile Neutropenia | After randomization until day 30
  Unique temperature >38.3°C or sustained temperature >38°C over the course of an hour, and a total count of neutrophils <1000 cells/mm3.

SECONDARY OUTCOMES:
Time passed from cisplatin-based chemotherapy until the apparition of febrile neutropenia | After randomization until day 30
  Total of days passed from the randomization up to the apparition of febrile neutropenia
Safety of Oral Supplementation with Magnesium | Evaluate the apparition of adverse effects of oral supplement of magnesium oxide Time Frame: After randomization until day 30
  Evaluate the apparition of adverse effects of oral supplement of magnesium oxide
Hypomagnesemia | After randomization until day 30
  Serum magnesium <1.6 mg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo D Castelán, PhD, Principal Investigator — Universidad Nacional Autónoma de México. Facultad de Estudios Superiores Zaragoza; Miguel A Palomo, PhD, Principal Investigator — Hospital Infantil de México Dr. Federico Gómez
Locations (1):
- Hospital Infantil de Mexico Dr. Federico Gomez, Cuauhtémoc, Mexico City, Mexico

REFERENCES:
- [Background] Freifeld AG, Pizzo PA. The outpatient management of febrile neutropenia in cancer patients. Oncology (Williston Park). 1996 Apr;10(4):599-606, 611-2; discussion 615-6. PMID 8723296
- [Background] Castagnola E, Paola D, Giacchino R, Rossi R, Viscoli C. Economic aspects of empiric antibiotic therapy for febrile neutropenia in children with cancer. Support Care Cancer. 1998 Nov;6(6):524-8. doi: 10.1007/s005200050208. PMID 9833301
- [Background] Mueller EL, Sabbatini A, Gebremariam A, Mody R, Sung L, Macy ML. Why pediatric patients with cancer visit the emergency department: United States, 2006-2010. Pediatr Blood Cancer. 2015 Mar;62(3):490-5. doi: 10.1002/pbc.25288. Epub 2014 Oct 24. PMID 25345994
- [Background] Klaassen RJ, Goodman TR, Pham B, Doyle JJ. "Low-risk" prediction rule for pediatric oncology patients presenting with fever and neutropenia. J Clin Oncol. 2000 Mar;18(5):1012-9. doi: 10.1200/JCO.2000.18.5.1012. PMID 10694551
- [Background] Castelan-Martinez OD, Rodriguez-Islas F, Vargas-Neri JL, Palomo-Colli MA, Lopez-Aguilar E, Clark P, Castaneda-Hernandez G, Rivas-Ruiz R. Risk Factors for Febrile Neutropenia in Children With Solid Tumors Treated With Cisplatin-based Chemotherapy. J Pediatr Hematol Oncol. 2016 Apr;38(3):191-6. doi: 10.1097/MPH.0000000000000515. PMID 26907640
- [Background] Lajer H, Daugaard G. Cisplatin and hypomagnesemia. Cancer Treat Rev. 1999 Feb;25(1):47-58. doi: 10.1053/ctrv.1999.0097. PMID 10212589
- [Background] Knijnenburg SL, Mulder RL, Schouten-Van Meeteren AY, Bokenkamp A, Blufpand H, van Dulmen-den Broeder E, Veening MA, Kremer LC, Jaspers MW. Early and late renal adverse effects after potentially nephrotoxic treatment for childhood cancer. Cochrane Database Syst Rev. 2013 Oct 8;(10):CD008944. doi: 10.1002/14651858.CD008944.pub2. PMID 24101439
- [Background] Willox JC, McAllister EJ, Sangster G, Kaye SB. Effects of magnesium supplementation in testicular cancer patients receiving cis-platin: a randomised trial. Br J Cancer. 1986 Jul;54(1):19-23. doi: 10.1038/bjc.1986.147. PMID 3524645
- [Background] Martin M, Diaz-Rubio E, Casado A, Lopez Vega JM, Sastre J, Almenarez J. Intravenous and oral magnesium supplementations in the prophylaxis of cisplatin-induced hypomagnesemia. Results of a controlled trial. Am J Clin Oncol. 1992 Aug;15(4):348-51. doi: 10.1097/00000421-199208000-00016. PMID 1514533
- [Background] Zarif Yeganeh M, Vakili M, Shahriari-Ahmadi A, Nojomi M. Effect of Oral Magnesium Oxide Supplementation on Cisplatin-Induced Hypomagnesemia in Cancer Patients: A Randomized Controlled Trial. Iran J Public Health. 2016 Jan;45(1):54-62. PMID 27057522
- [Derived] Castelan-Martinez OD, Palomo-Colli MA, Barrios-Lopez VE, Silva-Jivaja KM, Juarez-Villegas LE, Castaneda-Hernandez G, Sanchez-Rodriguez MA. Efficacy and safety of oral magnesium supplementation in reducing febrile neutropenia episodes in children with solid tumors treated with cisplatin-based chemotherapy: randomized clinical trial. Cancer Chemother Pharmacol. 2020 Nov;86(5):673-679. doi: 10.1007/s00280-020-04155-4. Epub 2020 Oct 8. PMID 33030582

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT03449693/Prot_SAP_002.pdf